CLINICAL TRIAL: NCT06281847
Title: An Adaptive Open-label Multicentre Phase 1/2 Trial, to Determine the Recommended Phase 2 Dose of CCTx-001, and to Assess Safety, Tolerability, and Clinical Activity in Patients With Relapsed/Refractory Acute Myeloid Leukaemia
Acronym: RESOLVE AML001
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Advesya SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCTx-001-AML-001
Record Dates: First submitted 2024-02-06; First posted 2024-02-28 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia, in Relapse; Acute Myeloid Leukemia Refractory
Keywords: Acute Myeloid Leukemia; Relapsed; Refractory; Open-label; Safety; Tolerability
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Intervention Model Description: The study comprises 4 periods:
  * The pre-treatment period will consist of screening for eligibility, leukapheresis and a pre-treatment evaluation (prior to Lymphodepleting Chemotherapy (LDC)).
  * The treatment period will start with LDC, followed by CCTx-001 infusion 2 to 7 days after completion of LDC. A first response evaluation will be performed at approximately 28 days after CCTx-001 infusion.
  * The post-treatment period will consist of further clinical activity and safety follow-up visits at regular timepoints after CCTx-001 infusion, starting after the Month 3 visit up to the Month 24 visit.
  * The long-term follow-up period will start after the Month 24 visit up to 15 years post CCTx-001 infusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label CCTx-001 infusion (Experimental): CCTx-001 infusion 2 to 7 days after completion of LDC
  Interventions: Genetic: CCTx-001

INTERVENTIONS:
Genetic: CCTx-001 — Frozen CAR T-cells suspensions in media containing dimethyl sulfoxide (DMSO)

SUMMARY:
The purpose of this adaptive Phase 1/2 study is to evaluate the safety, tolerability, pharmacokinetics (PK), and antileukemic activity of CCTx-001 in adult patients with r/r Acute Myeloid Leukemia (AML). CCTx-001 targets IL-1RAP, which is specifically expressed in leukemic cells. In preclinical studies, IL-1RAP-targeted Chimeric antigen receptors (CARs) have demonstrated encouraging activity in both in vitro and in vivo experiments in AML models. Based on these promising preclinical results, it is expected that CCTx-001 could potentially alter the natural course of r/r AML and provide a potential novel treatment option.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with active (> 5 % blasts in bone marrow) r/r AML (WHO 2022) who have exhausted their therapeutic alternatives or have contraindications to these alternatives as judged by the treating physician defined as either:

   a. Primary refractory: i. Patients who failed after two cycles of intensive induction including high-dose and/or standard dose cytarabine (including liposomal formulation), +/- anthracycline, +/- antimetabolite, +/- targeted therapy or ii. Older patients or patients unfit to receive intensive induction courses who failed after two cycles of venetoclax + azacitidine or 4 cycles of azacitidine b. Relapsing: i. Patients with early relapse after CR to first line therapy (within ≤ 6 months after CR1) or ii. Patients with relapse after later lines of therapy (Relapse after CR≥2) c. Patients relapsing after allogeneic hematopoietic stem cell transplant: i. Patients must be at least 3 months from hematopoietic stem cell transplant (HSCT) at the time of consent, and ii. Off immunosuppression for at least 1 month at the time of consent, and iii. Have no active graft versus host disease (GvHD)
2. Have a circulating blast count of less than 20,000/mm3 (control with hydroxyurea is allowed)
3. Absolute Lymphocyte count of >200/mm3
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
5. Life expectancy of more than 3 months
6. Patient is ≥ 18 years of age at the time of informed consent
7. Read, understood, and signed the informed consent form (ICF) prior to any study procedures
8. Patient is willing and able to adhere to the study visit schedule and other protocol requirements
9. Eligible for leukapheresis
10. Treatment-related toxicities of previous therapies have completely resolved
11. Adequate organ function as confirmed by clinical laboratory values, defined as:

    1. Adequate bone marrow function to receive LDC as assessed by the Investigator
    2. Serum creatinine [< 1.5 x the upper limit of normal (ULN) or creatinine clearance (CrCl) > 45 mL/min] (estimated by Cockcroft Gault or Modification of Diet in Renal Disease (MDRD); see Appendix 14.3 for calculation)
    3. Alanine aminotransferase [≤ 3 x ULN and total bilirubin < 1.5 mg/dL (or < 3.0 mg/dL] for patients with Gilbert's syndrome or leukemic infiltration of the liver)]
    4. Adequate pulmonary function, defined as [≤ Grade 1 dyspnoea according to CTCAE and oxygen saturation (SaO2) ≥ 92% on room air and forced expiratory volume in the first second ≥ 50%]
    5. Ejection fraction > 40% assessed by an echocardiogram (ECHO) or multigated acquisition (MUGA) scan performed within 1 month before CCTx-001 infusion
12. Women of childbearing potential* (WOCBP) must have a negative serum pregnancy test performed at screening and within 7 days before enrolment
13. WOCBP or males whose sexual partners are WOCBP must be able and willing to use at least 1 highly effective method of contraception during the study and for 12 months after the last dose of LDC. For the definition and list of highly effective methods of contraception.

Exclusion Criteria:

1. Patients with an acute promyelocytic leukaemia: t(15;17)(q22;q12); (promyelocytic leukaemia/retinoic acid receptor alpha) and variants
2. Patients with active central nervous system (CNS) leukaemia involvement. If the patient has prior history of CNS leukaemia, they must have a negative cerebrospinal fluid (CSF) assessment and magnetic resonance imaging (MRI) or computed tomography (if MRI is not feasible) of the brain demonstrating no evidence of CNS disease
3. Patients with isolated extramedullary AML disease
4. Patients who received previous treatment targeting IL-1RAP or previous gene therapy
5. Patients who underwent allo-HSCT within 90 days prior to leukapheresis
6. Patients who received donor lymphocyte infusion within 60 days prior to leukapheresis
7. Patients with active GvHD
8. Patients with history of another primary malignancy other than disease under study unless the patient has been free of the disease for ≥ 2 years, except for the following non-invasive malignancies:

   1. Basal cell carcinoma of the skin
   2. Squamous cell carcinoma of the skin
   3. Carcinoma in situ of the cervix
   4. Carcinoma in situ of the breast
   5. Incidental histologic finding of prostate cancer (T1a or T1b) or prostate cancer that is curative
   6. Other completely resected stage 1 solid tumour with low risk for recurrence
9. Presence of systemic fungal, bacterial, viral, or other infection (including tuberculosis) that is uncontrolled despite appropriate antibiotics or other treatments
10. Active or prior history of hepatitis B or hepatitis C infection
11. History of or active human immunodeficiency virus (HIV) infection
12. Active macrophage activation syndrome (MAS) as evidenced by laboratory abnormalities (e.g.: elevated ferritin, elevated triglycerides, haemophagocytosis on the bone marrow sample) and/or clinical signs
13. History or presence of an active and clinically relevant CNS disorder such as epilepsy, generalised seizure disorder, paresis, aphasia, stroke, cerebral oedema, severe brain injury, dementia, multiple sclerosis, Parkinson's disease, cerebellar disease, organic brain syndrome, or posterior reversible encephalopathy syndrome, or any autoimmune disease with CNS involvement
14. Patients with active autoimmune disorders or active neurological or inflammatory disorders (e.g., Guillain-Barre Syndrome, Amyotrophic Lateral Sclerosis) requiring immunosuppressive therapy or corticosteroid therapy (defined as >20 mg/day prednisone or equivalent). Physiologic replacement, topical, and inhaled steroids are permitted.
15. Use of the following (see Section 8.3 for full details):

    1. Therapeutic doses of corticosteroids (defined as > 20 mg/day prednisone or equivalent) within 7 days prior to leukapheresis or 72 hours prior to CCTx-001 infusion. Physiologic replacement, topical, and inhaled steroids are permitted.
    2. Immunosuppressive therapies within 4 weeks prior to signing the ICF (e.g., calcineurin inhibitors, methotrexate or other chemotherapeutics, mycophenolate, rapamycin, thalidomide, immunosuppressive antibodies such as anti-tumour necrosis factor [TNF], anti-IL-6, or anti-IL-6 receptor [IL-6R])
    3. Cytotoxic chemotherapeutic agents (including intrathecal) within 14 days prior to leukapheresis.
    4. Treatment with alemtuzumab within 6 months of leukapheresis, or treatment with fludarabine or cladribine within 3 months of leukapheresis
    5. Experimental agents within 4 weeks prior to signing the ICF unless no response or progressive disease (PD) is documented on the experimental therapy and at least 3 half-lives have elapsed prior to signing the ICF.
    6. Therapeutic anticoagulation
16. History of any one of the following cardiovascular conditions within the past 6 months prior to signing the ICF:

    1. Class III or IV heart failure as defined by the New York Heart Association
    2. Cardiac angioplasty or stenting
    3. Myocardial infarction
    4. Unstable angina
    5. Other clinically significant cardiac disease
17. Known hypersensitivity to DMSO or other excipients
18. Uncontrolled medical, psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol, as judged by the Investigator; or unwillingness or inability to follow the procedures required in the protocol.
19. Abnormal findings and/or clinically significant Grade ≥3 non-haematological toxicity and any other medical condition(s) or laboratory findings that, in the opinion of the Investigator, might jeopardise the patient's safety.
20. Presence of any condition that confounds the ability to interpret data from the study based on Investigator´s judgement.
21. Any planned medical/surgical treatment that might interfere with the ability to comply with the study requirements.
22. Pregnant or nursing women. NOTE: WOCBP must have a negative serum pregnancy test performed within 48 hours of starting LDC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2041-08 (Estimated)

PRIMARY OUTCOMES:
Phase 1: To evaluate the safety, tolerability, and to define the recommended phase 2 dose (RP2D) of CCTx-001 | Up to 28 days
  Frequency, severity, relationship and persistence of adverse events (AEs) and dose-limiting toxicity (DLTs)
Phase 2: To evaluate the clinical activity, as assessed by the composite complete response rate, in patients treated with CCTx-001 | Up to 3 months
  Composite complete response rate (cCRR) defined as the proportion of patients with best overall response, as assessed by Independent Review Committee (IRC) based on European LeukemiaNet (ELN) 2022 criteria, at complete remission (CR), CR with partial haematologic recovery (CRh), or CR with incomplete haematologic recovery (CRi).

SECONDARY OUTCOMES:
Phase 2: To evaluate the clinical activity, as assessed by the complete remission rate, in patients treated with CCTx-001 | Up to 3 months
  Complete remission rate (CRR) defined as the proportion of patients with best overall response, as assessed by IRC based on ELN 2022 criteria, at CR.
Phase 1: To evaluate the clinical activity, as assessed by the composite complete response rate, in patients treated with CCTx-001 | Up to 3 months
  cCRR
Phase 2: To assess the safety of CCTx-001 | Up to 15 years
  Frequency, severity, relationship and persistence of AEs
Phase 1 & 2: To assess additional parameters of clinical activity in patients treated with CCTx-001 | Up to 3 months
  Objective response rate (ORR)
Phase 1 & 2: To assess additional parameters of clinical activity in patients treated with CCTx-001 | Up to 24 months
  event-free survival (EFS)
Phase 1 & 2: To assess additional parameters of clinical activity in patients treated with CCTx-001 | Up to 24 months
  relapse-free survival (RFS)
Phase 1 & 2: To assess additional parameters of clinical activity in patients treated with CCTx-001 | Up to 15 years
  overall survival (OS)
Phase 1 & 2: To assess additional parameters of clinical activity in patients treated with CCTx-001 | Up to 24 months
  duration of response (DOR)
Phase 1 & 2: To assess additional parameters of clinical activity in patients treated with CCTx-001 | Up to 24 months
  cumulative incidence of relapse (CIR)
Phase 1 & 2: To assess additional parameters of clinical activity in patients treated with CCTx-001 | Up to 24 months
  cumulative incidence of death (CID)
Phase 1 & 2: To assess additional parameters of clinical activity in patients treated with CCTx-001 | Up to 24 months
  time to composite complete response (TTcCR)
Phase 1 & 2: To assess additional parameters of clinical activity in patients treated with CCTx-001 | Up to 3 months
  time to response (TTR) according to ELN 2022 criteria and minimal residual disease (MRD) responses
Phase 1 & 2: To evaluate the overall safety and the tolerability of CCTx-001 | Up to 15 years
  Frequency and severity of AEs and laboratory abnormalities

CONTACTS AND LOCATIONS:
Locations (6):
- France (2):
  - Besançon Regional and University Hospital, Besançon
  - Hospital Saint Louis, Paris
- Germany (2):
  - Ludwig-Maximilians University of Munich, Munich
  - University Hospital Ulm, Ulm
- Vall d'Hebron University Hospital, Barcelona, Spain
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No